CLINICAL TRIAL: NCT00971035
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study to Evaluate Lebrikizumab (MILR1444A) in Adult Patients With Asthma Who Are Not Taking Inhaled Corticosteroids (MOLLY)
Brief Title: A Study to Evaluate Lebrikizumab (MILR1444A) in Adult Patients With Asthma Who Are Not Taking Inhaled Corticosteroids
Acronym: MOLLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILR4660g
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: MILR1444A
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Experimental)
  Interventions: Drug: lebrikizumab (MILR1444A)
- B (Experimental)
  Interventions: Drug: lebrikizumab (MILR1444A)
- C (Experimental)
  Interventions: Drug: lebrikizumab (MILR1444A)
- D (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lebrikizumab (MILR1444A) — Subcutaneous repeating dose
  Arms: A
Drug: lebrikizumab (MILR1444A) — Subcutaneous repeating dose
  Arms: B
Drug: lebrikizumab (MILR1444A) — Subcutaneous repeating dose
  Arms: C
Drug: placebo — Subcutaneous repeating dose
  Arms: D

SUMMARY:
This is a randomized, double-blind, placebo controlled, four-arm, dose-ranging study. The purpose is to evaluate the relationship between the dose of lebrikizumab and the response in terms of the efficacy, safety, and tolerability in patients with asthma who are not on inhaled steroids.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 50 kg and ≤ 150 kg at Visit 1
* Chest radiograph within 12 months of Visit 1 without evidence of a clinically significant abnormality
* Stable asthma

Exclusion Criteria:

* Asthma exacerbation during screening
* Known malignancy
* Known immunodeficiency
* Pre-existing lung disease other than asthma
* Uncontrolled clinically significant medical disease
* Current smoker
* History of substance abuse that may impair or risk the patient's full participation in the study, in the judgment of the investigator
* Prior allergic reaction to a monoclonal antibody
* Patients (men and women) of reproductive potential who are not willing to use contraception
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in 1 second (FEV1) | Baseline to Week 12

SECONDARY OUTCOMES:
Change in pre-bronchodilator FEV1 | Baseline to Week 24
Change in quality of life and symptom scores | Baseline to Week 12
Change in peak flow | Baseline to Week 1
Rate of asthma exacerbations | During the 24-week treatment period
Change in rescue medication use | From baseline to Week 1
Frequency and severity of adverse events | From the first study-specific procedure through the last observation visit
Incidence of human anti-therapeutic antibodies (ATA) | Baseline to Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Freemer, M.D., Study Director — Genentech, Inc.